CLINICAL TRIAL: NCT04848207
Title: Effect of Open Tray Versus Digital Impressions on the Passivity and Prosthetic Complications of Full Arch Screw-retained Prosthesis - A Randomized Control Trial Study
Brief Title: Effect of Open Tray Versus Digital Impressions on the Passivity and Prosthetic Complications of Full Arch Screw-retained Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Hassan Hussein Mohamed Elsharkawy, MSc faculty of Dentistry, Cairo university (2019), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO 6-2-2
Record Dates: First submitted 2021-04-06; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Passivity; Prosthetic Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital impression technique (Other): - 3D printed generic Scan bodies with unified shape and length replacing the traditional transfer copings will be press fitted on the trans-mucosal abutments and pickup cylinders that are screwed on the implants to capture their position and intra-oral scanning will be done.
  Interventions: Device: Digital impression technique
- Open tray impression technique (Other): * Transfer copings will be screwed to the multiunit abutments on the existing implants, and splinted together using pre-cured printed resin splinting framework that will be fixed to the copings using flowable composite .
  * A one step impression technique using putty and light addition silicon will be made, where light impression material will be injected all around transfer copings and putty silicon will be loaded in tray and then will be seated intra-orally making sure to fully expose the screws of transfer copings through the impression material.
  Interventions: Other: Open tray impression technique

INTERVENTIONS:
Device: Digital impression technique — 3D printed generic Scan bodies with unified shape and length replacing the traditional transfer copings will be press fitted on the trans-mucosal abutments and pickup cylinders that are screwed on the implants to capture their position and intra-oral scanning will be done.
  Arms: Digital impression technique
Other: Open tray impression technique — Transfer copings will be screwed to the multiunit abutments on the existing implants, and splinted together using pre-cured printed resin splinting framework that will be fixed to the copings using flowable composite .
  A one step impression technique using putty and light addition silicon will be made, where light impression material will be injected all around transfer copings and putty silicon will be loaded in tray and then will be seated intra-orally making sure to fully expose the screws of transfer copings through the impression material.
  Arms: Open tray impression technique

SUMMARY:
The importance of this trial lies in testing if intraoral digital impressions will increase the accuracy of impressions of full arch implant cases over conventional impression techniques thus improving the passivity of full arch screw retained prosthesis and decreasing the prosthetic complications in turn.

DETAILED DESCRIPTION:
In this study intraoral digital impressions will be used for scanning full arch implant cases to minimize the variables in the conventional technique, finally the study will investigate if the intraoral digital impressions will increase the accuracy of impressions of full arch implant cases thus improving the passivity and decreasing prosthetic complications of screw retained prosthesis for a long-term success compared to open tray impression technique.

Primary outcome will be evaluation of the passivity of PMMA (Polymethyl methacrylate ) try-in , while secondary outcomes will be detecting prosthetic complications (screw loosening , prosthesis fracture) and treatment time for both groups.

Eligibility criteria:

Inclusion criteria:

* Completely edentulous patients with sufficient inter-arch space to receive fixed prosthesis (Crown height space 9-15 mm per arch)
* Completely edentulous patients with 4 implants in mandible and/ or 6 implants in maxilla
* sufficient bone volume for implant placement without graft a confirmed by CBCT
* adequate zone of keratinized mucosa ( > 2mm width)
* All genders
* Acceptable oral hygiene
* Cooperative patients
* Controlled systemic diseases ( Diabetes, hypertension)

Exclusion criteria:

* Completely edentulous patients with insufficient inter-arch space to receive fixed prosthesis ( Crown height space lesser than 9mm per arch)
* Insufficient bone volume for implant placement
* Completely edentulous patients with in-adequate zone of keratinized mucosa (< 2mm).
* Un cooperative patients
* Poor oral hygiene
* Uncontrolled diabetic patients( Diabetes, hypertension)

Interventions:

Completely edentulous patients that have received dental implants and ready to start prosthetic steps of full arch screw retained prosthesis will be recruited and randomly divided into two groups.

Group 1 ( control group):

* Primary impression will be taken followed by customization of open special trays for each patient.
* Transfer copings will be screwed to the multiunit abutments on the existing implants, and splinted together using pre-cured printed resin splinting framework that will be fixed to the copings using flowable composite and one step impression technique using putty and light addition silicon will be made . Implant analogs will be attached to the transfer copings and pouring of the impression will be done using dental stone.
* Bite registration will be done followed by mounting of stone casts on the articulator.
* Patient's stone models and bite will be scanned using desktop scanner and the trial PMMA bridge will be designed and 3D-printed as a verification jig to evaluate the accuracy of the taken impression.
* Passivity of the trial PMMA bridge will be evaluated on patients intra-orally using single screw test, peri-apical radiographs and Screw resistance parameter (SR parameter).
* Regarding the final prosthesis a framework will be designed on the patient's scan and milled from (PEEK blocks) , finished and polished then layered by (pink composite ) and (composite teeth) will be used.
* Final prosthesis will be delivered to the patient and treatment time will be measured by the number of visits starting from impression taking session till delivery session.
* Follow up of the patients will be done every at 3 and 6 months to check if there are any prosthetic complications (screw loosening or fracture).

while in Group 2 ( intervention group):

* Intra-oral scanner will be used in the study to take a digital impression for the implants.
* 3D printed generic Scan bodies with unified shape and length replacing the traditional transfer copings will be press fitted on the trans-mucosal abutments and pickup cylinders that are screwed on the implants to capture their position and intra-oral scanning will be done.
* With scan bodies in place, bite will be registered where, in case of completely edentulous upper and lower arches a 3D printed centric holding device will be used to fix the vertical dimension at the desired height and the intra-oral scanner will capture the bite at this position, but in case of a completely edentulous arch opposed by dentulous arch , a green stick jig will be customized anteriorly to hold vertical dimension at the desired height and intra-oral scanner will be used to record the bite bilaterally.
* The STL file of the captured scan will be 3D-printed into a resin model with negative places replicating the analogues design in which the digital analogues will be seated.
* The trial PMMA bridge will be designed on the implants scan then 3D- printed, to be fitted on the resin model having digital analogues in place.
* Passivity of the trial PMMA bridge will be evaluated on patients the same way as group 1.
* The final prosthesis a framework will be designed and milled as in group 1 then delivered to the patient outcomes:
* Passivity of PMMA tryin: will be measured by Single screw test, Periapical radiograph, Screw resistance parameter (SR parameter) at PMMA tryin visit (2nd visit after impressions Instantly).
* Prosthetic complications (screw loosening , prosthesis fracture) : will be measured by Clinical examination at 3, 6 months of delivery of final prosthesis.
* Treatment time : will be measured by Number of visits at the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients with sufficient inter-arch space to receive fixed prosthesis (Crown height space 9-15 mm per arch)
* Completely edentulous patients with 4 implants in mandible and/ or 6 implants in maxilla
* sufficient bone volume for implant placement without graft a confirmed by CBCT
* adequate zone of keratinized mucosa ( > 2mm width)
* All genders
* Acceptable oral hygiene
* Cooperative patients
* Controlled systemic diseases ( Diabetes, hypertension)

Exclusion Criteria:

* Completely edentulous patients with sufficient inter-arch space to receive fixed prosthesis (Crown height space 9-15 mm per arch)

  * Completely edentulous patients with 4 implants in mandible and/ or 6 implants in maxilla
  * sufficient bone volume for implant placement without graft a confirmed by CBCT
  * adequate zone of keratinized mucosa ( > 2mm width)
  * All genders
  * Acceptable oral hygiene
  * Cooperative patients
  * Controlled systemic diseases ( Diabetes, hypertension)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Passivity of seating of PolyMethylMethAcrylate (PMMA) tryin prosthesis | 3-4 months after implants placement after final impressions for implants
  the screw retained prosthesis can be considered passive when it does not generate static loads and strains within the prosthesis or in the surrounding bone structure measured using Single screw test (measuring unit : binary - yes/No)
Passivity of seating of PolyMethylMethAcrylate (PMMA) tryin prosthesis | 3-4 months after implants placement after final impressions for implants
  the screw retained prosthesis can be considered passive when it does not generate static loads and strains within the prosthesis or in the surrounding bone structure measured using
  -Periapical radiograph ( measuring unit : binary- Yes/No)
Passivity of seating of PolyMethylMethAcrylate (PMMA) tryin prosthesis | 3-4 months after implants placement after final impressions for implants
  the screw retained prosthesis can be considered passive when it does not generate static loads and strains within the prosthesis or in the surrounding bone structure measured using
  - Screw resistance parameter (Measuring unit: Difference of rotation angles in passive and non- passive situations)

SECONDARY OUTCOMES:
Prosthetic complications including screw loosening and prosthesis fracture | At 3, 6 months after delivery of final prosthesis
  screw loosening , prosthesis fracture will be assessed by clinical examination (measuring unit : number of times )
Treatment time | 5-6 months after implants placement ( at the last visit )
  Number of visits

IPD SHARING:
Plan to Share IPD: No